CLINICAL TRIAL: NCT00520273
Title: A Prospective Study to Evaluate the Specificity of the Cobas TaqScreen MPX Test for Use on the Cobas s 201 System for Screening Plasma Pools From Source Plasma Donors for the Presence of HBV DNA, HCV RNA, and HIV-1 RNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000487; CAT-MPX-143
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Volunteer

ARMS (1):
- A (Experimental)
  Interventions: Device: cobas s 201 TaqScreen MPX Test

INTERVENTIONS:
Device: cobas s 201 TaqScreen MPX Test — Donors testing reactive for one or more of the viral markers will be advised to seek further advice/treatment from their physician.

SUMMARY:
This study will evaluate the specificity of the cobas TaqScreen MPX Test for the simultaneous detection of HBV DNA, HCV RNA and HIV-1 Group M in a minimum of 100,000 individual donor samples in 96-unit pools.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-65 years of age
* Fulfil criteria for plasma donation

Exclusion Criteria:

* Do not fulfil criteria for plasma donation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Source plasma donors were screened for the presence of HIV-1 RNA, HBV DNA, and/or HCV RNA | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Ziermann, Study Director — Roche Molecular Systems, Inc
Locations (3):
- United States (3):
  - Boca Raton, Florida
  - Raleigh, North Carolina
  - Memphis, Tennessee